CLINICAL TRIAL: NCT03457844
Title: A Single Group, Open Label, Multi-center Clinical Trial to Assess the Efficacy and Safety of Anlotinib in Patients With Gastroenteropancreatic Neuroendocrine Tumor G3
Brief Title: A Study of Anlotinib in Patients With Gastroenteropancreatic Neuroendocrine Tumor G3
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-13-II
Record Dates: First submitted 2018-02-27; First posted 2018-03-08 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-03

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumor G3
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib (Experimental)
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib is followed Day 1 to day 14 by 7 days off treatment in a 21-day cycle） and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent

SUMMARY:
To assess the primary effects and safety of Anlotinib in patients with Gastroenteropancreatic Neuroendocrine Tumor G3.

ELIGIBILITY:
Inclusion Criteria:

* Patients should participate in the study voluntarily and sign informed consent;
* 18-75 years old;
* Histopathological proven diagnosis of high grade (G3) advanced Gastroenteropancreatic Neuroendocrine Tumor(Unresectable locally advanced or distant Metastatic). the classification is based on the Ki-67 proliferative index >20%(WHO 2010),and Provision of qualified pathological tissue for central review;
* Progression during or after treatment with first-line systematic chemotherapy;
* At least one measurable nidus (by RECIST1.1);
* Main organs function is normal;
* Eastern Cooperative Oncology Group(ECOG) performance status(PS):0-1,Life expectancy of more than 12 weeks;
* Women of childbearing potential should agree to use and utilize an adequate method of contraception (such as intrauterine device，contraceptive and condom) throughout treatment and for at least 6 months after study is stopped；the result of serum or urine pregnancy test should be negative within 7 days prior to study enrollment，and the patients required to be non-lactating；Man participants should agree to use and utilize an adequate method of contraception throughout treatment and for at least 6 months after study is stopped;

Exclusion Criteria:

* Diagnosed with low or intermediate (G1,G2) neuroendocrine tumors, Manec, adenocarcinoma;
* Functional neuroendocrine tumors(NETs) which need to be treated with long acting somatostatin analogue(SSAs) to control disease related syndromes, such as insulinoma, gastrinoma, glucagonoma, somatostatinoma, accompanied by carcinoid syndrome, Zollinger-Ellison syndrome or other active symptoms;
* Other malignancies diagnosed within the previous 5 years, except basal cell carcinoma or cervical carcinoma in situ after radical resection；
* Have received anti-vascular endothelial growth factor（VEGF）/VEGFR targeted drugs and progressed upon these drugs；
* Patients with factors that could affect oral medication (such as dysphagia，chronic diarrhea, intestinal obstruction etc.)
* Patients with any severe and/or unable to control diseases，including：

  1. Blood pressure unable to be controlled ideally(systolic pressure≥150 mmHg，diastolic pressure≥100 mmHg);
  2. Patients with Grade 1 or higher myocardial ischemia, myocardial infarction or malignant arrhythmias(including QT≥480ms) and patients with Grade 1 or higher congestive heart failure (NYHA Classification);
  3. Patients with active or unable to control serious infections;
  4. Patients with cirrhosis, decompensated liver disease, or active hepatitis;
  5. Patients with poorly controlled diabetes (fasting blood glucose(FBG)>10mmol/L)
  6. Urine protein ≥ ++，and 24-hour urinary protein excretion>1.0g confirmed;
* Patients had surgery (except biopsy) within 28 days or the surgical incision has not fully healed before the first study drug implementation;
* Patients with brain metastasis or spinal cord compression which had not surgical and / or radiation therapy,or which had previous treatment but there is no clinical imaging evidence proving the condition is stable;
* Anti-tumor therapy was performed within 4 weeks prior to initiation of the study treatment, including but not limited to chemotherapy, radical radiotherapy, bio-targeted therapy, immunotherapy, anti-tumor treatment of traditional Chinese medicine, hepatic artery embolization, hepatic metastatic cryoablation or radiofrequency ablation surgery.Palliative radiotherapy for a bone metastasis lesion within 2 weeks prior to the initiation of the investigational treatment;
* The toxic reaction of previous anticancer treatment has not been restored to grade 0 or 1 (except hair loss);
* Patients with arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism;
* Imaging showed tumors have involved important blood vessels or by investigators determine likely during the follow-up study and cause fatal hemorrhage;
* Patients with drug abuse history and unable to get rid of or Patients with mental disorders;
* Patients participated in other anticancer drug clinical trials within 4 weeks;
* History of immunodeficiency;
* Pregnancy(Positive detection of pregnancy before drug use)or lactation;
* Patients with concomitant diseases which could seriously endanger their own safety or could affect completion of the study according to investigators' judgment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival(PFS) | From randomization，each 42 days up to progressive disease(PD) or death(up to 24 months)

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
Overall survival(OS) | From randomization until death (up to 24 months)
Disease Control Rate(DCR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Yihebali Chi, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No